CLINICAL TRIAL: NCT02166970
Title: Single Versus Multiple Deployment of Metallic Stents for Inoperable Malignant Hilar Biliary Obstruction: A Multicenter Prospective Randomized Study
Brief Title: Single Versus Multiple Deployment of Metallic Stents for Inoperable Malignant Hilar Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae Hoon Lee, Professor, Soon Chun Hyang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hilar stenting
Record Dates: First submitted 2014-06-13; First posted 2014-06-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Klatskin Tumor
Keywords: Hilar tumor; Metal stent; Single; Multiple
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single stent deployment (Experimental): Metallic stent deployment in hilar obstruction. Insertion of metallic stent to the dominant targeted duct such as right anterior (segments V and VIII), right posterior (segments VI and VII) or left (segments II-IV).
  Interventions: Device: Metallic stent deployment in hilar obstruction
- Multiple stent deployment (Active Comparator): Metallic stent deployment in hilar obstruction. Insertion of multiple metallic stent to the dominant targeted duct such as right anterior (segments V and VIII), right posterior (segments VI and VII) or left (segments II-IV).
  Interventions: Device: Metallic stent deployment in hilar obstruction

INTERVENTIONS:
Device: Metallic stent deployment in hilar obstruction — Single stent insertion: metal stent deployment to right or left intrahepatic duct Multiple stenting: Stent-in-stent or side-by-side deployment
  Other Names: Single stent insertion; Multiple stent insertion using stent-in-stent method; Multiple stent insertion using side-by-side method

SUMMARY:
In Bismuth II-IV hilar cholangiocarcinoma patients with a predicted survival of longer than 3 months, metallic stent performance is superior to plastic stenting for palliation with respect to outcomes and cost-effectiveness. However, the optimal stent type and the extent of drainage are issues that remain to be definitively decided. The optimal endoscopic management strategy is contentious. The investigators conduct the present study to prospectively in multi-centers compare unilateral (single) with bilateral (multiple) deployment in inoperable malignant biliary obstructions to clarify the clinical outcomes of these two deployment methods using metallic stents.

DETAILED DESCRIPTION:
In Bismuth II-IV hilar cholangiocarcinoma patients with a predicted survival of longer than 3 months, metallic stent performance is superior to plastic stenting for palliation with respect to outcomes and cost-effectiveness.

However, the optimal stent type and the extent of drainage are issues that remain to be definitively decided. The optimal endoscopic management strategy is contentious.

The investigators conduct the present study to prospectively in multi-centers compare unilateral (single) with bilateral (multiple) deployment in inoperable malignant biliary obstructions to clarify the clinical outcomes of these two deployment methods using metallic stents.

First as an unilateral or bilateral stent will be deployed according to criteria.

In bilateral group, stent-in-stent or side-by-side deployment will be included.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* inoperable hilar malignancy

Exclusion Criteria:

* age under 18 years
* uncontrolled coagulopathy
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Reintervention rate when stents occluded | 2 years
  When the stents occluded after successful single or multiple stent deployment, the outcome measure is assessed.

SECONDARY OUTCOMES:
Technical success of single or multiple stents | 1 month
  When the bilirubin level decrease more than 50% within one week or 75% within one month.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hoon Lee, MD, PhD, Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Tae Hoon Lee, Cheonan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee TH, Kim TH, Moon JH, Lee SH, Choi HJ, Hwangbo Y, Hyun JJ, Choi JH, Jeong S, Kim JH, Park DH, Han JH, Park SH. Bilateral versus unilateral placement of metal stents for inoperable high-grade malignant hilar biliary strictures: a multicenter, prospective, randomized study (with video). Gastrointest Endosc. 2017 Nov;86(5):817-827. doi: 10.1016/j.gie.2017.04.037. Epub 2017 May 4. PMID 28479493